CLINICAL TRIAL: NCT02429284
Title: United States CTEPH Registry
Brief Title: U.S. CTEPH Registry
Status: Completed | Type: Observational
Sponsor: University of California, San Diego (Other)
Collaborators: E Squared Trials and Registries, Inc. (Industry)
Responsible Party: Principal Investigator, Kim Kerr, Clinical Professor of Medicine, University of California, San Diego
Other Study IDs: PH-2013-008
Record Dates: First submitted 2015-04-13; First posted 2015-04-29 (Estimated); Last update posted 2020-03-24 (Actual); Status verified 2020-03

CONDITIONS: Chronic Thromboembolic Pulmonary Hypertension (CTEPH); Pulmonary Hypertension
Keywords: Chronic Thromboembolic Pulmonary Hypertension (CTEPH); Pulmonary Endarterectomy (PEA); Pulmonary Thromboendarterectomy (PTE); Pulmonary Hypertension; Balloon Pulmonary Angioplasty (BPA)
MeSH Terms: conditions — Hypertension, Pulmonary

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 4 Years
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Patients newly diagnosed with CTEPH: Patients newly diagnosed with chronic thromboembolic pulmonary hypertension (CTEPH), WHO Group IV Classification for Pulmonary Hypertension.

SUMMARY:
The U.S. CTEPH Registry is a multicenter, observational, U.S.-based study of the clinical course and treatment of patients diagnosed with chronic thromboembolic pulmonary hypertension (CTEPH), WHO Group IV Classification for Pulmonary Hypertension. The mission of the Registry will be to promote a greater understanding of the prevalence, pathophysiology, evaluation, and treatment of patients with CTEPH through shared information, education, and collaborative investigation among pulmonary hypertension (PH) centers of excellence throughout the U.S.

DETAILED DESCRIPTION:
Chronic thromboembolic pulmonary hypertension (CTEPH) is a subset of pulmonary hypertension (PH) characterized by the obstruction of pulmonary arteries with fibrotic material and vascular remodeling that leads to increased pulmonary arterial pressure and right ventricular failure.

A United States CTEPH Registry has been established under the guidance of a Steering Committee consisting of recognized physicians and scientists with expertise in CTEPH and related diseases. The mission of the Registry will be to promote a greater understanding of the prevalence, pathophysiology, evaluation, and treatment of patients with CTEPH through shared information, education, and collaborative investigation among PH centers of excellence throughout the U.S. The development of a national CTEPH registry will be an important element in the advancement of the understanding of CTEPH and improvement in the care of patients who suffer from this debilitating disease.

All consecutive consenting patients recently diagnosed (< 6 months) with CTEPH at participating study sites will be enrolled. At the time of study entry, data on prior history and evaluation will be obtained from patient interview and review of medical records. Patients will be followed biannually after enrollment until the conclusion of the study (minimum of 1 year follow-up for final patients enrolled).

Much of the data gathered by the Registry will be presented as descriptive statistics. The Registry will seek the assistance of a biostatistician to develop a statistical plan for within patient and between patient cohort analyses.

Approximately 750 patients with newly diagnosed (< 6 months) CTEPH will be enrolled.

TIME FRAME:

Participants will be followed from the time of their enrollment until 1 year after the final patient is enrolled. Short term outcome measures and medical history will be collected during the initial visit, and clinical data will be collected from the initial clinic visits, hospital says, or procedures (if applicable). Patients will then be followed every 6 months after their enrollment for long term outcome measures on quality of life, functional status, and medical treatments.

DATA ANALYSES:

Demographics and Clinical Course:

Demographics, risk factors, time to appropriate testing and diagnosis, PAH targeted medication use, functional status, and hemodynamics at the time of enrollment will be provided annually as aggregate data to all investigators.

Evaluating Outcomes of PTE Surgery:

Descriptive statistics of the peri-operative data collected will be provided as aggregate data to all investigators annually. Immediate post-operative and longitudinal follow-up of all patients undergoing PTE surgery will also be provided as aggregate data annually to all sites. Comparisons of hemodynamics, functional status, medication and supplemental oxygen use and healthcare utilization will be made between the pre-operative data and longitudinal post-operative data.

Evaluating Predictors of Successful PTE:

Using longitudinal data collected on post-operative PTE patients, a definition of "successful PTE" will be established based upon hemodynamics, functional status and QoL. Retrospective analysis of pre-, peri-, and post-operative data can then be analyzed to identify factors that predict a "successful" or "unsuccessful" PTE surgery.

Evaluating Outcomes of Nonsurgical Therapy of CTEPH:

Predominantly descriptive statistics will be used to describe why patients are not operative candidates and the nonsurgical therapies (medication, balloon pulmonary angioplasty) used for treatment. Changes in hemodynamics, functional status, QoL and healthcare utilization on therapy will be provided as aggregate data annually.

Evolving Research Needs:

To adapt to the evolving science and research needs of the CTEPH community, separate analysis plans will be developed for new objectives identified and minor changes in the eCRF may occur in response to new diagnostics and treatments, if approved by the Steering Committee. Ongoing assessment of enrollment and data captured will also be performed by the Steering Committee to be certain the goals of the Registry are being met.

COMMITTEES:

A Steering Committee, chaired by Dr. Kim Kerr, is comprised of thought leaders in the areas of cardiology, pulmonology, and cardiothoracic surgery with expertise in CTEPH. The committee will have the following responsibilities:

* Provide advice and guidance on the U.S. CTEPH Registry study design and protocol
* Provide advice and guidance on the variables to be captured by the eCRF
* Provide guidance on study sites selection
* Review data results and provide insights into interpretation of the data annually
* Provide input on the planning and organization of abstracts and manuscripts
* Review abstracts and papers for submission to scientific journals or conferences
* Present data at conferences

An Adjudication Committee, consisting of physicians with expertise in the diagnosis of CTEPH, will review all patients felt by Investigators to be eligible for the Registry. The adjudication committee members must confirm the diagnosis of CTEPH before the subject can be enrolled in the Registry.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be a permanent resident of the United States
* Documentation of the following hemodynamic parameters by right heart catheterization

  * Mean pulmonary arterial pressure (PAPm) ≥ 25 mm Hg at rest and,
  * Pulmonary artery wedge pressure (PAWP) ≤ 15 mm Hg (or > 15 mmHg if justified)
* Radiologic confirmation that chronic thromboembolic disease is the cause of the pulmonary hypertension by

  * One or more mismatched perfusion defect(s) by lung ventilation/perfusion scan, and
  * Confirmation of chronic thromboembolic disease by evidence of bands/webs, vessel narrowing or occlusion seen on CT pulmonary angiogram (CTA), conventional angiography or MR angiography (MRA).
* Patients must be diagnosed with CTEPH within 6 months of being considered for study eligibility (signing of consent to participate). The date of diagnosis will be defined as when both hemodynamic criteria have been met and chronic thromboembolic disease is confirmed to be the cause of the pulmonary hypertension by an abnormal V/Q scan and the presence of chronic thromboembolic disease on CTA, MRA or pulmonary angiography. Hemodynamic and radiologic criteria can be met at separate time points; the most recently met criteria time point will be defined as the date of diagnosis.
* Prior to enrollment all subjects must have the diagnosis of CTEPH confirmed by the Adjudication Committee.

Exclusion Criteria:

* Patients unwilling or unable to provide written consent for participation in the study. Appropriate surrogate consent will be obtained for pediatric patients as defined by each investigational site's IRB.
* Patients with an underlying medical disorder with an anticipated life expectancy less than 2 years.
* Patients who do not meet inclusion criteria including:

  * Have not had documentation of hemodynamic criteria by right heart catheterization as outlined in the inclusion criteria
  * Do not have radiologic confirmation of chronic thromboembolic disease as outlined in the inclusion criteria
  * Meet the criteria for inclusion into WHO Groups I, II, III, or V

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All consecutive consenting patients recently diagnosed (< 6 months) with CTEPH at participating study sites will be enrolled. Patients must meet inclusion criteria and have the diagnosis of CTEPH confirmed by the Adjudication Committee (AC) to be enrolled. Adult and pediatric patients may be enrolled and prior medical therapy will not exclude patients from enrollment.
Sampling Method: Non-Probability Sample
Enrollment: 754 (Actual)
Dates: Start 2015-04 (Actual); Primary Completion 2019-05 (Actual); Study Completion 2019-11 (Actual)

PRIMARY OUTCOMES:
Describe the patterns of evaluation of CTEPH Patients | up to 5 years
Describe the patters of risk factors and clinical presentation of CTEPH Patients | up to 5 years
Outcomes of medical and surgical therapy of CTEPH patients as assessed by hemodynamics, quality of life, and functional status | up to 5 years, at 6 month intervals

CONTACTS AND LOCATIONS:
Overall Officials: Kim M Kerr, MD, Principal Investigator — University of California, San Diego
Locations (1):
- UCSD Health System, La Jolla, California, United States

REFERENCES:
- [Background] Kim NH, Delcroix M, Jenkins DP, Channick R, Dartevelle P, Jansa P, Lang I, Madani MM, Ogino H, Pengo V, Mayer E. Chronic thromboembolic pulmonary hypertension. J Am Coll Cardiol. 2013 Dec 24;62(25 Suppl):D92-9. doi: 10.1016/j.jacc.2013.10.024. PMID 24355646
- [Background] McGoon MD, Benza RL, Escribano-Subias P, Jiang X, Miller DP, Peacock AJ, Pepke-Zaba J, Pulido T, Rich S, Rosenkranz S, Suissa S, Humbert M. Pulmonary arterial hypertension: epidemiology and registries. J Am Coll Cardiol. 2013 Dec 24;62(25 Suppl):D51-9. doi: 10.1016/j.jacc.2013.10.023. PMID 24355642
- [Background] Pepke-Zaba J, Delcroix M, Lang I, Mayer E, Jansa P, Ambroz D, Treacy C, D'Armini AM, Morsolini M, Snijder R, Bresser P, Torbicki A, Kristensen B, Lewczuk J, Simkova I, Barbera JA, de Perrot M, Hoeper MM, Gaine S, Speich R, Gomez-Sanchez MA, Kovacs G, Hamid AM, Jais X, Simonneau G. Chronic thromboembolic pulmonary hypertension (CTEPH): results from an international prospective registry. Circulation. 2011 Nov 1;124(18):1973-81. doi: 10.1161/CIRCULATIONAHA.110.015008. Epub 2011 Oct 3. PMID 21969018
- [Derived] Kerr KM, Elliott CG, Chin K, Benza RL, Channick RN, Davis RD, He F, LaCroix A, Madani MM, McLaughlin VV, Park M, Robbins IM, Tapson VF, Terry JR, Test VJ, Jain S, Auger WR. Results From the United States Chronic Thromboembolic Pulmonary Hypertension Registry: Enrollment Characteristics and 1-Year Follow-up. Chest. 2021 Nov;160(5):1822-1831. doi: 10.1016/j.chest.2021.05.052. Epub 2021 Jun 4. PMID 34090871
- [Derived] Kerr KM, Elliott CG, Benza RL, Channick RN, Chin KM, Davis RD, Jain S, LaCroix AZ, Madani MM, McLaughlin VV, Park MH, Tapson VF, Auger WR. The United States Chronic Thromboembolic Pulmonary Hypertension Registry: Protocol for a Prospective, Longitudinal Study. JMIR Res Protoc. 2021 May 25;10(5):e25397. doi: 10.2196/25397. PMID 33848258